CLINICAL TRIAL: NCT07139132
Title: Transforming Risk Factors in a High Stroke Risk Native American Population Through a Cultural Nutritional Program
Brief Title: The AHA Oneida Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American Heart Association (AHA) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-1171; SMPH/NEURO SURG/NEURO SURG (Other: UW Madison); FA (Other: UW Madison); Protocol Version 10/2/25 (Other: UW Madison)
Record Dates: First submitted 2025-08-12; First posted 2025-08-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Oneida Nation Members
MeSH Terms: interventions — Ultrasonography, Carotid Arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- School-age Native Americans (Experimental): Participants who are age 7-17 and live with adult parent or guardian will answer a 10 question nutritional knowledge questionnaire.
  Interventions: Behavioral: Health Wellness Coaching; Diagnostic Test: Carotid ultrasound; Behavioral: School-age nutritional education program; Diagnostic Test: Cognitive Testing
- Adult Native Americans (Experimental): Adults age 18-85
  Interventions: Behavioral: Health Wellness Coaching; Diagnostic Test: Carotid ultrasound; Diagnostic Test: Cognitive Testing; Diagnostic Test: Blood work

INTERVENTIONS:
Behavioral: Health Wellness Coaching — Health wellness coach will provide education and guidance about cultural nutrition
Diagnostic Test: Carotid ultrasound — Participants will undergo an ultrasound
Behavioral: School-age nutritional education program — Educational program will teach students about healthy Native American food choices
  Arms: School-age Native Americans
Diagnostic Test: Cognitive Testing — Participants will undergo a cognitive test.
Diagnostic Test: Blood work — Participants will undergo blood work.
  Arms: Adult Native Americans

SUMMARY:
The purpose of this clinical trial is to learn whether a cultural nutritional program can change stroke risk factors, cognitive decline, and learn how school education programs about nutrition can improve health in the Oneida Nation.

Participants will undergo:

* A carotid ultrasound
* Cognitive testing
* Health assessment
* Blood work
* Health wellness coaching

Participants can expect to be in the study for 1 year.

DETAILED DESCRIPTION:
The specific aims for this study are: 1) to determine if a cultural nutritional program across generations can change stroke risk factors in the Oneida Nation; 2) to determine if a cultural nutritional program across generations can change vascular cognitive decline in the Oneida Nation; and, 3) determine how structured culturally competent school education programs about nutrition influence knowledge of health. The intervention used is health wellness coaching. All individuals enrolled in this study will have opportunity to interact with an Oneida Nation employed Health wellness coach to find out about Oneida resources that they can use to modify their stroke risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-85 years
* Receiving healthcare though the Oneida Comprehensive Health Division

Exclusion Criteria:

* Not Native American

Ages: 7 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in incidence of stroke and transient ischemic attack (TIA) | Baseline to 1 year
  Number of incidences of stroke or TIA during the study
Change in number of participants that meet American Heart Association (AHA) Simple Rules for Diastolic Blood Pressure. | Baseline to 1 year
  The AHA's simple rules for diastolic blood pressure: Normal = Less than 80 mm Hg; Elevated = Less than 80 mm Hg with a systolic reading of 120-129 mm Hg; Stage 1 Hypertension = 80-89 mm Hg; Stage 2 Hypertension = 90 mm Hg or higher; Hypertensive Crisis = Higher than 120 mm Hg (along with a systolic reading higher than 180 mm Hg). Researchers will be reporting the change in number of participants with diastolic blood pressure <90 mmHg.
Change in number of participants that meet AHA's Simple Rules for Systolic Blood Pressure. | Baseline to 1 year
  The AHA uses these simple rules for systolic blood pressure (the top number): Normal is less than 120, Elevated is 120-129, Stage 1 Hypertension is 130-139, and Stage 2 Hypertension is 140 or higher. A systolic reading of 180 or higher indicates a hypertensive emergency. Researchers will be reporting the change in number of participants with systolic blood pressure <140 mmHg.
Change in number of participants that meet AHA Simple Rules for Body Mass Index (BMI) | Baseline to 1 year
  The AHA uses the following guidelines for Body Mass Index (BMI) in adults:
  Underweight = Less than 18.5; Normal Weight = Between 18.5 and 24.9; Overweight = Between 25 and 29.9; and, Obesity = 30 or higher. Researchers will be reporting any improvement in BMI.
Change in Montreal Cognitive Assessment (MoCA) | Baseline to 1 year
  MoCA is scored out of a total of 30 points, with a score of 26 or above generally considered normal. The MoCA assesses various cognitive domains, including memory, visuospatial abilities, language, and executive functions. A lower score indicates potential cognitive impairment, with specific cutoffs for mild (19-23), moderate (10-18), and severe (0-9) impairment.
Change in NIH Toolbox Score | Baseline to 1 year
  NIH Toolbox Cognition Battery consists of tests of multiple constructs to asses for cognitive, sensory, motor and emotional function
Change in Native American Acculturation Scale (NAAS) | Baseline to 1 year
  NAAS is a 20-item questionnaire developed to assess the level of acculturation in Native Americans. It measures an individual's connection to both traditional Native American culture and mainstream American culture. Scores range from a low of 1, indicating low acculturation (or high Native American identity) to a high of 5, indicating high acculturation (or high mainstream American identity), with a score of 3 indicating "bicultural". The NAAS examines areas like identity, language, friendships, behaviors, attitudes, and generational/geographic background.
Change in knowledge of health through a structured culturally competent school education programs about nutrition | Baseline to 1 year

SECONDARY OUTCOMES:
Change in nutrition knowledge | Baseline to 1 year
  Change in knowledge will be assessed with pre-test, 1 year post-test of each participant to assess improvement in nutritional knowledge and understanding of healthy food options tied to Oneida culture. This will be assessed through a 10-question multiple choice survey about good versus bad nutrition choices. Participants will select their choices, low score indicates poor nutritional knowledge and high score indicating better understanding for healthy nutrition
Change in plaque area | Baseline to 1 year
  Measured via carotid ultrasound.
Change in pulsatility index in carotid arteries | Baseline to 1 year
  Measured via carotid ultrasound. This index is a unitless measurement calculated: peak systolic velocity - end diastolic velocity, divided by the mean velocity, higher values are thought to represent increased resistance to blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dempsey, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Oneida Nation Reservation, Oneida, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes